CLINICAL TRIAL: NCT06914102
Title: Emulation of the STEP-HFpEF DM Heart Failure Trial in Healthcare Claims Data
Acronym: DUP-STEP-HFpEF
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-STEP-HFpEF
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2; HFpEF - Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Semaglutide: Exposure group
  Interventions: Drug: Semaglutide
- Placebo: Reference group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — New use of semaglutide dispensing claim is used as the exposure.
  Groups: Semaglutide
Drug: Placebo — New use of sitagliptin dispensing claim is used as the reference (active-comparator proxy for placebo).
  Groups: Placebo

SUMMARY:
Investigators are building an empirical evidence base for real-world data through large-scale emulation of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the Randomized Controlled Trials Duplicated Using Prospective Longitudinal Insurance Claims: Applying Techniques of Epidemiology (RCT DUPLICATE) initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to emulate, as closely as is possible in healthcare insurance claims data, the STEP-HFpEF DM trial described below. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. In addition to closely emulating the trial population, this study also evaluates outcomes in a broader, less restrictive cohort to enhance generalizability to patients typically encountered in routine clinical practice.

Randomization cannot be achieved in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides guidance on the reference standard treatment effect estimate. However, failure to replicate RCT findings is not necessarily indicative of the inadequacy of the healthcare claims data for emulation for a range of possible reasons, as the end points examined in the database study were only of exploratory nature in the trial. Moreover, divergence from these end points do not provide information on the validity of the original RCT finding.

The STEP-HFpEF DM trial is a superiority trial that included an evaluation of the effect of semaglutide, a glucagon-like peptide-1 receptor agonist (GLP-1-RA), vs placebo on all-cause mortality or worsening heart failure events among individuals with heart failure with preserved ejection fraction.

The database study designed to emulate STEP-HFpEF DM will be a new-user active-comparative study, conducted using 3 national United States claims databases, where we compare the effect of semaglutide vs sitagliptin, a dipeptidyl peptidase-4 inhibitor (DPP4i) on the composite end point of all-cause mortality or heart failure hospitalization. While the STEP-HFpEF DM trial compared semaglutide vs placebo, we chose to use sitagliptin as an active-comparator proxy for placebo. Sitagliptin was specifically chosen because a major randomized controlled trial on cardiovascular outcomes demonstrated that the drug does not affect the cardiovascular outcomes under investigation. Furthermore, clinical guidelines during the study period recommended both drug classes under investigation as second- or third-line options for glucose lowering and were similarly costly

ELIGIBILITY:
Eligible cohort entry dates:

Optum: Study period between January 1, 2018 to November 30, 2024. Marketscan: Study period between January 1, 2018 to December 31, 2023. Medicare: Study period between January 1, 2018 to December 31, 2020.

FOLLOWING ELIGIBILITY OF THE STEP-HFpEF DM TRIAL

Inclusion Criteria:

* Male or female, age above or equal to 18 years at the time of signing informed consent.
* BMI ≥ 30.0 kg/m2
* NYHA Class II-IV
* LVEF ≥ 45%
* No hospitalizations due to heart failure between screening (V1) and randomization (V2)
* At least one of the following:
* If BMI <35.0: NT-proBNP ≥ 220 pg/mL (for patients with sinus rhythm) or NTproBNP ≥660 pg/mL (for patients with persistent/permanent atrial fibrillation); if BMI ≥ 35.0: NT-proBNP ≥ 125 pg/mL (for patients with sinus rhythm) or NTproBNP ≥ 375 pg/mL (for patients with persistent/permanent atrial fibrillation) at screening (NT-proBNP analyzed by the central laboratory) in combination with at least one of the following (documented by echocardiography within 12 months prior to or at screening): i. Septal é < 7cm/sec or lateral é < 10 cm/sec or average E/é ≥ 15 ii. PA systolic pressure >35mmHg iii. Left atrial (LA) enlargement (LA width ≥3.8 cm or LA length ≥ 5.0cm or LA area ≥ 20.0cm2 or LA volume ≥ 55mL or LA volume index ≥29mL/m2) iv. LV hypertrophy with septal thickness or posterior wall thickness ≥1.2cm
* Hospitalization with a primary diagnosis of decompensated heart failure which required intravenous loop diuretic treatment, within the previous 12 months in combination with at least two of the following (documented by echocardiography within 12 months prior to or at screening): i. Septal é < 7cm/sec or lateral é < 10cm/sec or average E/é ≥15 ii. PA systolic pressure >35mmHg iii. LA enlargement (LA width ≥3.8cm or LA length ≥ 5.0cm or LA area ≥20.0cm2 or LA volume ≥ 55mL or LA volume index ≥ 29mL/m2) iv. LV hypertrophy with septal thickness or posterior wall thickness ≥1.2cm
* Diagnosed with T2D ≥ 90 days prior to the day of screening.
* Subject treated with diet, exercise, and/or antidiabetic treatment* according to local label in stable dosing for at least 30 days prior to screening: o *OAD(s): unchanged drug(s), dose and dosing frequency o *Insulin(s): unchanged regimen (basal, basal + bolus, premix combination) with stable total daily insulin dose as judged by the investigator

Exclusion Criteria:

* Myocardial infarction, stroke, hospitalization for heart failure, unstable angina pectoris or transient ischemic attack within 30 days prior to the day of screening.
* Systolic blood pressure > 160 mmHg at screening.
* Any other condition judged by the investigator to be the primary cause of dyspnea (such as heart failure due to restrictive cardiomyopathy or infiltrative conditions (e.g. amyloidosis), hypertrophic obstructive cardiomyopathy, primary pulmonary arterial hypertension, chronic obstructive pulmonary disease, right heart failure due to pulmonary disease, complex congenital heart disease, anemia, or more than moderate heart valve disease).
* Bariatric surgery prior to screening or planned bariatric surgery within the trial time course.
* History of type 1 diabetes (history of gestational diabetes is allowed).
* Treatment with any GLP-1 receptor agonist within 90 days prior to the day of screening.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy.
* Recurrent severe hypoglycemic episodes within the last year as judged by the investigator.
* Treatment with continuous subcutaneous insulin infusion
* Personal or first-degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma.
* Presence of acute pancreatitis within the last 180 days prior to screening.
* History or presence of chronic pancreatitis.
* End-stage renal disease or chronic or intermittent hemodialysis or peritoneal dialysis.
* Presence or history of malignant neoplasm within 5 years prior to the day of screening. Basal and squamous cell cancer and any carcinoma in-situ are allowed.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method.
* Any disorder, including severe psychiatric disorder, suicidal behavior within 90 days before screening, and suspected drug abuse, which in the investigator´s opinion might jeopardize subject´s safety or compliance with the protocol.

RELAXING ELIGIBILITY OF THE STEP-HFpEF DM TRIAL

Inclusion Criteria:

* Men or women ≥ 18 years old
* History of type 2 diabetes mellitus
* BMI ≥ 27.0 kg/m2
* Heart failure
* Preserved ejection fraction

Exclusion Criteria:

* Prior treatment with any GLP-1-RA
* History of type 1 diabetes mellitus
* End-stage renal disease or chronic or intermittent hemodialysis or peritoneal dialysis
* History of bariatric surgery
* History of nursing home admission
* Pregnant female or breast-feeding
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy
* Treatment with continuous subcutaneous insulin infusion
* Multiple endocrine neoplasia type 2 or medullary thyroid carcinoma
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy (other than basal- or squamous-cell skin cancer, in situ carcinoma of the cervix, or in situ prostate cancer) for less than 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population included individuals aged 18 years or older with heart failure with preserved ejection fraction when following and relaxing the eligibility criteria of the STEP-HFpEF DM trial.
Sampling Method: Non-Probability Sample
Enrollment: 58387 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality or heart failure hospitalization | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of semgalutide vs placebo (sitaglitpin) on composite of all-cause mortality or heart failure hospitalization in two populations (1) patients meeting the eligibility criteria of the STEP-HFpEF DM trial, and (2) a broader patient population when relaxing the eligibility criteria of the STEP-HFpEF DM trial.

SECONDARY OUTCOMES:
Composite of all-cause mortality or a worsening heart failure event (exacerbated symptoms of heart failure resulting in hospitalization, intravenous diuretic therapy in an urgent care setting), and its respective individual end points. | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of semgalutide vs placebo (sitaglitpin) on composite of all-cause mortality or all-cause mortality or a worsening heart failure event (exacerbated symptoms of heart failure resulting in hospitalization, intravenous diuretic therapy in an urgent care setting) in two populations (1) patients meeting the eligibility criteria of the STEP-HFpEF DM trial, and (2) a broader patient population when relaxing the eligibility criteria of the STEP-HFpEF DM trial.
Worsening heart failure event (exacerbated symptoms of heart failure resulting in hospitalization or intravenous diuretic therapy in an urgent care setting) | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of semgalutide vs placebo (sitaglitpin) on worsening heart failure event (exacerbated symptoms of heart failure resulting in hospitalization or intravenous diuretic therapy in an urgent care setting) in two populations (1) patients meeting the eligibility criteria of the STEP-HFpEF DM trial, and (2) a broader patient population when relaxing the eligibility criteria of the STEP-HFpEF DM trial.
Intravenous diuretic therapy in an urgent care setting | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of semgalutide vs placebo (sitaglitpin) on intravenous diuretic therapy in an urgent care setting in two populations (1) patients meeting the eligibility criteria of the STEP-HFpEF DM trial, and (2) a broader patient population when relaxing the eligibility criteria of the STEP-HFpEF DM trial.
Hospitalization for heart failure | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of semgalutide vs placebo (sitaglitpin) on hospitalization for heart failure in two populations (1) patients meeting the eligibility criteria of the STEP-HFpEF DM trial, and (2) a broader patient population when relaxing the eligibility criteria of the STEP-HFpEF DM trial.
All-cause mortality | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of semgalutide vs placebo (sitaglitpin) on all-cause mortality in two populations (1) patients meeting the eligibility criteria of the STEP-HFpEF DM trial, and (2) a broader patient population when relaxing the eligibility criteria of the STEP-HFpEF DM trial.
Urinary tract infection | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of semgalutide vs placebo (sitaglitpin) on urinary tract infection in two populations (1) patients meeting the eligibility criteria of the STEP-HFpEF DM trial, and (2) a broader patient population when relaxing the eligibility criteria of the STEP-HFpEF DM trial.
Serious bacterial infection | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of semgalutide vs placebo (sitaglitpin) on serious bacterial infection in two populations (1) patients meeting the eligibility criteria of the STEP-HFpEF DM trial, and (2) a broader patient population when relaxing the eligibility criteria of the STEP-HFpEF DM trial.
Gastrointestinal adverse events | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of semaglutide vs placebo (sitagliptin) on gastrointestinal adverse events in two populations: (1) patients meeting the eligibility criteria of the STEP-HFpEF DM trial, and (2) a broader patient population when relaxing the eligibility criteria of the STEP-HFpEF DM trial.

OTHER OUTCOMES:
Hernia | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of semaglutide vs placebo (sitagliptin) on a negative control outcome of hernia in two populations: (1) patients meeting the eligibility criteria of the STEP-HFpEF DM trial, and (2) a broader patient population when relaxing the eligibility criteria of the STEP-HFpEF DM trial.
Lumbar radiculopathy | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of semaglutide vs placebo (sitagliptin) on a negative control outcome of lumbar radiculopathy in two populations: (1) patients meeting the eligibility criteria of the STEP-HFpEF DM trial, and (2) a broader patient population when relaxing the eligibility criteria of the STEP-HFpEF DM trial.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital; Nils Krüger, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kruger N, Schneeweiss S, Fuse K, Matseyko S, Sreedhara SK, Hahn G, Schunkert H, Wang SV. Semaglutide and Tirzepatide in Patients With Heart Failure With Preserved Ejection Fraction. JAMA. 2025 Oct 14;334(14):1255-1266. doi: 10.1001/jama.2025.14092. PMID 40886075

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT06914102/Prot_SAP_001.pdf